CLINICAL TRIAL: NCT02293161
Title: A Randomised, Double-Blind (Sponsor Unblind), Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of Single Ascending Doses of a Fully Humanized Anti-IL-7 Receptor α Monoclonal Antibody (GSK2618960) in Healthy Volunteers
Brief Title: Single Ascending Doses Study of Anti- Interleukin-7 Receptor α Monoclonal Antibody (GSK2618960) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200902
Record Dates: First submitted 2014-10-27; First posted 2014-11-18 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Autoimmune Diseases
Keywords: Interleukin-7 Receptor α; monoclonal antibody
MeSH Terms: conditions — Autoimmune Diseases | interventions — GSK2618960

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A GSK2618960 (Experimental): Subjects will receive GSK2618960 0.6 milligram per kilogram (mg/kg)
  Interventions: Drug: GSK2618960
- Cohort A Placebo (Placebo Comparator): Subjects will receive Sodium Chloride Intravenous as placebo
  Interventions: Drug: Placebo
- Cohort B GSK2618960 (Experimental): Subjects will receive GSK2618960,planned dose being 2mg/kg. However, actual dose level for Cohort B may be adjusted based on the emerging data on safety, tolerability, PK and RO from Cohort A. The maximum dose will not exceed 2.4 mg/kg (i.e. a 4-fold dose escalation from 0.6 mg/kg)
  Interventions: Drug: GSK2618960
- Cohort B Placebo (Placebo Comparator): Subjects will receive Sodium Chloride Intravenous as placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2618960 — GSK2618960 will be provided as 100 mg/mL solution for injection to be administered as single dose IV infusion that has to be diluted at the study site with placebo
  Arms: Cohort A GSK2618960; Cohort B GSK2618960
Drug: Placebo — It is Sodium Chloride Intravenous Infusion
  Arms: Cohort A Placebo; Cohort B Placebo

SUMMARY:
GSK2618960 is a humanized Immunoglobulin G 1 ( IgG1) monoclonal antibody (mAb) that binds to the alpha component (CD127) of the heterodimeric Interleukin-7 receptor (IL-7R). It is being developed for the treatment of autoimmune indications. This study is intended to further explore the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of single ascending doses GSK2618960 in healthy volunteers beyond those already evaluated in I7R116702 (First Time In Human study). The study is anticipated to enrol 18 subjects in total, with 9 subjects in each of the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 18 and 65 years of age inclusive, at the time of signing the informed consent OR females of non-child bearing potential aged between 18 and 65 years of age at the time of signing the informed consent.

Non-childbearing potential defined as:- pre-menopausal females with a documented tubal ligation or hysterectomy, or post-menopausal defined as 24 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli-international units (MIU) per millilitre (mL) and oestradiol <40 picograms (pg) /mL (< 140 picomole/liter) is confirmatory. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt must discontinue HRT to allow confirmation of postmenopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their postmenopausal status, they can resume use of HRT during the study.]

* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Protocol. This criterion must be followed from the time of the first dose of study medication until 5 half-lives after the infusion (Week 16 visit).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinically significant abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the local reference range being used for healthy volunteers may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* White blood cell count >=Lower Limit of Normal (LLN), including both lymphocyte and neutrophil counts >=LLN.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 19.0 - 32.0 kilogram / square meter (kg/m^2) (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subjects with a confirmed positive vaccination status for tetanus, diphtheria, pertussis, measles, mumps, rubella, pneumococcus and meningococcus (or consent to vaccination)

Exclusion Criteria:

Criteria Based Upon Medical Histories

* Current evidence of ongoing or acute infection within 3 months prior to the first dose of study drug, such as: serious local infection (e.g. cellulitis, abscess); systemic infection [e.g. pneumonia, septicaemia, Tuberculosis (TB)].
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A QT duration corrected for heart rate by Fridericia's formula (QTcF) >450 millisecond (msec) based on either single or averaged QTcF values of triplicate ECGs obtained over a brief recording period.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint ~240 mL of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Previous history of anaphylaxis and severe allergic reaction.
* Receipt of live vaccination within 1 month of screening or plan to receive live vaccination at any time during the study i.e. 6 months following dosing (which covers the period when the predicted target duration of receptor occupancy is >= 95%).
* Subjects from a high risk area of the world for tuberculosis or have history of tuberculosis or have close family members with confirmed TB infection or positive at screening by Quantiferon testing (an indeterminate test result at screen may be repeated once).

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface and/or core antibody or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody. Other Criteria
* Smokers who would not be able to refrain from smoking whilst in the phase I unit.
* Unable to refrain from the use of prescription or non-prescription drugs (unless permitted as per protocol
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day "rolling" period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse events (AE) | Up to Day 169
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Absolute values of vital signs | Up to Day 169
  Vital signs includes systolic and diastolic blood pressure, pulse rate and body temperature.
Change from baseline in vital signs | Baseline (Day1) and up to Day 169
  Vital signs includes systolic and diastolic blood pressure, pulse rate and body temperature.
Absolute values of Electrocardiogram (ECG) parameters | Up to Day 169
  Single 12-lead ECGs will be obtained.
Change from baseline in ECG parameters | Baseline (Day1) and up to Day 169
  Single 12-lead ECGs will be obtained.
Absolute values of haematology | Up to Day 169
  Haematology parameters includes Platelet Count, Red blood cells (RBC) Count, White blood cells Count (absolute) (WBC), Haemoglobin and Haematocrit
Change from baseline in haematology | Baseline (Day -1) and up to Day 169
  Haematology parameters includes Platelet Count, RBC, WBC, Haemoglobin and Haematocrit
Absolute values of clinical chemistry | Up to Day 169
  Clinical chemistry includes Blood urea nitrogen, Potassium, Aspartate aminotransferase (SGOT), Total and direct bilirubin, Creatinine, Chloride, Alanine aminotransferase (SGPT), Albumin, Glucose, Total Carbon dioxide, Gamma glutamyltransferase, Total Protein, Sodium, Calcium and Alkaline phosphatase
Change from baseline in clinical chemistry | Baseline (Day -1) and up to Day 169
  Clinical chemistry includes Blood urea nitrogen, Potassium, SGOT, Total and direct bilirubin, Creatinine, Chloride, SGPT, Albumin, Glucose, Total Carbon dioxide, Gamma glutamyltransferase, Total Protein, Sodium, Calcium and Alkaline phosphatase
Absolute values of urinalysis | Up to Day 169
  Urinalysis includes Specific gravity, pH, glucose, protein, blood and ketones by dipstick, Microscopic examination (if blood or protein is abnormal)
Change from baseline in urinalysis | Baseline (Day -1) and up to Day 169
  Urinalysis includes Specific gravity, pH, glucose, protein, blood and ketones by dipstick, Microscopic examination (if blood or protein is abnormal)

SECONDARY OUTCOMES:
Composite of PK parameters | Up to Day 29
  PK parameters includes Area Under the Concentration-time curve (AUC) from zero (pre-dose) extrapolated to infinite time (AUC[0-infinite]); AUC from time zero (pre-dose) to last quantifiable concentration within a subject across all treatments (AUC[0-t]); Percentage of AUC(0- infinite) obtained by extrapolation (%AUC-[ex]); Clearance (CL); Volume of distribution (Vss); Maximum observed concentration (Cmax); Time of occurrence of Cmax (Tmax); Terminal half life (t1/2).
Duration of full receptor occupancy (RO) for Cohort A | Up to Day 43
  The extent and duration of receptor occupancy and the inhibition of IL-7 signalling in Stat5 phosphorylation (pSTAT5) will be determined
Duration of full RO for Cohort B | Up to Day 57
  The extent and duration of receptor occupancy and the inhibition of IL-7 signalling in pSTAT5 will be determined
Relationship between dose/exposure and duration of full RO for Cohort A | Up to Day 43
  The PD/RO relationship of GSK2618960 following single and repeat Intravenous (IV) doses will be determined.
Relationship between dose/exposure and duration of full RO for Cohort B | Up to Day 57
  The PD/RO relationship of GSK2618960 following single and repeat IV doses will be determined.
Degree of blocking of IL-7R alpha signalling for Cohort A | Up to Day 43
  It will be assessed by residual IL-7- and Thymic Stromal Lymphopoietin (TSLP)-mediated pSTAT5 and Thymus and Activation-Regulated Chemokine (TARC) secretion
Degree of blocking of IL-7R alpha signalling for Cohort B | Up to Day 57
  It will be assessed by residual IL-7- and TSLP-mediated pSTAT5 and TARC secretion
Incidence of anti-drug antibodies (ADAs) | Up to Day 85
  Blood samples will be collected for the assessment of ADAs in serum using validated electrochemiluminescent (ECL)assays
Titre of ADAs | Up to Day 85
  Blood samples will be collected for the assessment of ADAs in serum using validated ECL assays

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- [Derived] Ellis J, van Maurik A, Fortunato L, Gisbert S, Chen K, Schwartz A, McHugh S, Want A, Santos Franco S, Oliveira JJ, Price J, Coles A, Brown K, Su D, Craigen JL, Yang J, Brett S, Davis B, Cheriyan J, Kousin-Ezewu O, Gray F, Thompson PW, Fernando D. Anti-IL-7 receptor alpha monoclonal antibody (GSK2618960) in healthy subjects - a randomized, double-blind, placebo-controlled study. Br J Clin Pharmacol. 2019 Feb;85(2):304-315. doi: 10.1111/bcp.13748. Epub 2018 Dec 3. PMID 30161291
- See also: Results for study 200902 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200902?search=study&b'study_ids=200902'#rs